CLINICAL TRIAL: NCT05508503
Title: Validation of a ctDNA Methylation-based Dual-target Test for the Detection of Colorectal Cancer: a Multicenter Clinical Study
Brief Title: A Study on a Blood-based Dual-target Test for CRC Detection
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); Qilu Hospital of Shandong University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, MD,Director, Head of Department of Gastroenterology and Digestive Endoscopy Center, Principal Investigator, Clinical Professor, Changhai Hospital
Other Study IDs: 2020CRC-cfDNA
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer; Colorectal Adenoma
Keywords: ctDNA; Methylation; Diagnostic test
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CRC group: patients with colorectal cancer
  Interventions: Diagnostic Test: Test of methylated NTMT1 and MAP3K14-AS1; Diagnostic Test: FIT
- Control group: patients without colorectal cancer
  Interventions: Diagnostic Test: Test of methylated NTMT1 and MAP3K14-AS1; Diagnostic Test: FIT

INTERVENTIONS:
Diagnostic Test: Test of methylated NTMT1 and MAP3K14-AS1 — A dual-target test kit to detect methylated NTMT1 and MAP3K14-AS1 in blood samples.
Diagnostic Test: FIT — Fecal immunochemical test（optional）

SUMMARY:
To evaluate the effectiveness and accuracy of the ctDNA dual-target test kit in a large case-control cohort for the detection of colorectal cancer and advanced adenomas.

DETAILED DESCRIPTION:
Usually, colorectal cancers (CRCs) diagnosed in their early stages are curable, especially precancerous lesions (adenomas, polyps) that can be removed during a colonoscopy.However, due to low patient compliance and limited resources, colonoscopy is not feasible for screening the average-risk population. gFOBT/FIT are limited by their low sensitivity and high false-positive rate. Compared to colonoscopy and stool DNA tests, blood-based methylation tests showed greater patient compliance and convenience. Hypermethylated NTMT1 and MAP3K14-AS1 were found in multiple cohorts of CRC samples in our previous study. In this study, we aimed to evaluate the effectiveness and accuracy of the ctDNA dual-target(NTMT1 and MAP3K14-AS1) test kit in 5 tertiary hospitals around china for the detection of colorectal cancer and advanced adenomas. Fecal immunochemical test (FIT) will also privided to participants in the study. Sanger sequencing would be performed to evalute the accuracy of the dual-target methylation detection test kit.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria for CRC group（≥30%） 1)Patients with colorectal cancer 2)Follow-up sample subjects: Subjects who underwent resection of colorectal cancer lesions.
2. Inclusion Criteria for Control group（≤70%） Health volunteer, or subject with other diseases or physiological conditions other than colorectal cancer, including but not limited to gastritis, gastric cancer, esophagitis, rheumatoid arthritis, prostate cancer, microbes (inflammation patients), gastrointestinal bleeding, drugs (typical digestive tract medication) Population), neuroendocrine cancer, squamous cell carcinoma (squamous squamous cell carcinoma, esophageal squamous cell carcinoma);

Exclusion Criteria:

1. Patients who had undergone radical resection of bowel cancer (except for postoperative follow-up) and those who had received anti-tumor therapy such as radiotherapy/chemotherapy；
2. Colorectal cancer or colorectal adenoma with other malignancies；
3. Postoperative follow-up patients of colorectal cance with distant metastasis;
4. The sample size collected did not meet the detection requirements;
5. Other patients who are considered unsuitable for this study (such as pregnancy, high blood pressure, heart disease, etc., who are not suitable for colonoscopy due to physical condition).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with colorectal cancer or subjects who referred to the outpatient and received colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 1378 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year.
  Sensitivity (for CRC and\or advanced precancerous neoplasm) of this blood-based methylation dual-target test. A diagnostic colonoscopy procedure is the reference method. Lesions will be confirmed as malignant or precancerous by histopathologic examination. Other clinically acceptable diagnostic criteria for non-intestinal diseases.
Specificity | Through study completion, an average of 1 year.
  Specificity (for CRC and\or advanced precancerous neoplasm) of this blood-based methylation dual-target test. A diagnostic colonoscopy procedure is the reference method. Lesions will be confirmed as malignant or precancerous by histopathologic examination. Other clinically acceptable diagnostic criteria for non-intestinal diseases.
Accuracy | Through study completion, an average of 1 year.
  Accuracy of the kit for methylation detection. Validation of the methylation status of MTNT1 and MAP3K14-AS1 by Sanger sequencing.

SECONDARY OUTCOMES:
Combined sensitivity | Through study completion, an average of 1 year.
  Sensitivity when combined the blood-based methylation dual-target test with FIT
Combined specificity | Through study completion, an average of 1 year.
  Specificity when combined the blood-based methylation dual-target test with FIT

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, MD, Principal Investigator — Changhai Hospital, Navy/Second Military Medical University
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Thierry AR, El Messaoudi S, Gahan PB, Anker P, Stroun M. Origins, structures, and functions of circulating DNA in oncology. Cancer Metastasis Rev. 2016 Sep;35(3):347-76. doi: 10.1007/s10555-016-9629-x. PMID 27392603
- [Background] Scholer LV, Reinert T, Orntoft MW, Kassentoft CG, Arnadottir SS, Vang S, Nordentoft I, Knudsen M, Lamy P, Andreasen D, Mortensen FV, Knudsen AR, Stribolt K, Sivesgaard K, Mouritzen P, Nielsen HJ, Laurberg S, Orntoft TF, Andersen CL. Clinical Implications of Monitoring Circulating Tumor DNA in Patients with Colorectal Cancer. Clin Cancer Res. 2017 Sep 15;23(18):5437-5445. doi: 10.1158/1078-0432.CCR-17-0510. Epub 2017 Jun 9. PMID 28600478
- [Background] Oster B, Thorsen K, Lamy P, Wojdacz TK, Hansen LL, Birkenkamp-Demtroder K, Sorensen KD, Laurberg S, Orntoft TF, Andersen CL. Identification and validation of highly frequent CpG island hypermethylation in colorectal adenomas and carcinomas. Int J Cancer. 2011 Dec 15;129(12):2855-66. doi: 10.1002/ijc.25951. Epub 2011 Apr 1. PMID 21400501
- [Background] Cao Y, Zhao G, Yuan M, Liu X, Ma Y, Cao Y, Miao B, Zhao S, Li D, Xiong S, Zheng M, Fei S. KCNQ5 and C9orf50 Methylation in Stool DNA for Early Detection of Colorectal Cancer. Front Oncol. 2021 Jan 29;10:621295. doi: 10.3389/fonc.2020.621295. eCollection 2020. PMID 33585248
- [Result] Chen H, Li N, Ren J, Feng X, Lyu Z, Wei L, Li X, Guo L, Zheng Z, Zou S, Zhang Y, Li J, Zhang K, Chen W, Dai M, He J; group of Cancer Screening Program in Urban China (CanSPUC). Participation and yield of a population-based colorectal cancer screening programme in China. Gut. 2019 Aug;68(8):1450-1457. doi: 10.1136/gutjnl-2018-317124. Epub 2018 Oct 30. PMID 30377193
- [Derived] Wang Z, He Z, Lin R, Feng Z, Li X, Sui X, Gu L, Xia T, Zhou D, Zhao B, Li Y, Li Z, Bai Y. Evaluation of a plasma cell-free DNA methylation test for colorectal cancer diagnosis: a multicenter clinical study. BMC Med. 2024 Oct 8;22(1):436. doi: 10.1186/s12916-024-03662-y. PMID 39379942